CLINICAL TRIAL: NCT02912767
Title: Prevalence of Self Reported Lymphedema in Patients With Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1001
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Endometrial Cancer; Lymphedema
Keywords: lower-extremity lymphedema; 16-1001
MeSH Terms: conditions — Endometrial Neoplasms; Lymphedema | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- SLN cohort: Patients who underwent hysterectomy only or with SLN mapping alone.
  Interventions: Behavioral: questionnaire
- LND cohort: Patients who underwent hysterectomy with standard lymphadenectomy, with or without SLN mapping.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — A questionnaire that has been validated by investigators at the Mayo Clinic. The questionnaire has 13 items to assess the rate of patient-reported lymphedema. The questionnaire will be mailed and then followed up with a second mailing after month 1 and a phone call after month 2. Within 3 months of sending the questionnaire a patient will be either considered as a responder vs non-responder. The date of surgery and the date of when the questionnaire is filled out will be captured.

SUMMARY:
The investigators are interested in understanding how the patient has been doing since their surgery for endometrial cancer and if they are experiencing any symptoms related to lymphedema (swelling) in the your lower body. The investigators hope that information from the patient and others will help them improve care for women treated for endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Presented to MSK with newly diagnosed endometrial carcinoma of any histologic profile clinically confined to the uterus and/or uterine cervix
* Underwent primary surgery at our institution, to include at least a total hysterectomy via laparotomy, laparoscopy, or robotic approach, between January 2006 and December 2013
* Alive at the time of study activation

Exclusion Criteria:

* Had documented macroscopic evidence of extrauterine disease at the time of initial diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from a retrospective database maintained by the GYN DMT. Patients will be contacted by mail for the first attempt at recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2016-07-20; Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
compare lymphedema prevalence | 1 year
  Data from respondents will be analyzed to determine prevalence of patient reported lymphedema overall; these will then be compared to the prevalence among those who underwent SLN mapping alone, or a comprehensive pelvic lymphadenectomy (+/- para-aortic LND and +/-SLN mapping in conjunction).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/